CLINICAL TRIAL: NCT06806683
Title: ITHACA: Development and Validation of a Multivariate Predictive Model for Prognosis in Head and Neck Cancer Patients Undergoing Radiotherapy - Ambispective Study.
Brief Title: Predictive Tools in Head and Neck Cancer Patients Undergoing Radiotherapy
Acronym: ITHACA
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6698
Record Dates: First submitted 2024-10-21; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancers; Head and Neck Cancers - Nasopharyngeal; Oral Cavity Cancer; Oropharyngeal Cancers; Radiotherapy Side Effects
Keywords: Head and neck cancer; Radiotherapy; Chemoradiotherapy; Radiomics; Personalized treatment; Dosiomics
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Oropharyngeal Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: intensity modulated radiotherapy — intensity modulated radiotherapy

SUMMARY:
The ITHACA study aims to improve the treatment of head and neck cancer by developing a predictive tool that helps doctors personalize care for each patient. This tool uses information such as medical history, imaging, and radiotherapy data to predict the risk of cancer recurrence, overall survival, and the likelihood of side effects.

Patients with head and neck cancer face significant challenges, including managing the side effects of treatments like radiotherapy. By tailoring treatment schedules and doses, and using advanced imaging techniques, we hope to reduce complications and improve survival outcomes. The study is designed to help doctors choose the best treatment for each patient, while minimizing the side effects that impact important functions like swallowing and breathing.

Patients participating in the study will have their medical data collected, including:

Tumor characteristics (size, location, stage). Treatment details (radiotherapy and chemotherapy). Imaging information using tools like PET-CT and MRI to track the response to treatment and detect any signs of cancer recurrence.

Side effects and overall health data. This information will be used to develop and test a new model that predicts outcomes for each patient based on their unique data.

The study includes adults (18 years and older) diagnosed with head and neck cancer, who are undergoing or have completed radiotherapy. Patients will be followed over time to monitor their response to treatment and any side effects.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria:

* Diagnosis: Confirmed head and neck cancer, including cancers of the oropharynx, larynx, hypopharynx, nasopharynx, salivary gland, unknown head and neck primary or oral cavity.
* Age: 18 years or older.
* Treatment: Undergoing or scheduled to undergo radiotherapy or chemoradiotherapy as part of their treatment

Exclusion Criteria

Participants will be excluded if they meet any of the following criteria:

* Pregnancy: Pregnant or breastfeeding women.
* Non-Compliance: Patients unwilling or unable to comply with study procedures and follow-ups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients (≥18 years old) diagnosed with head and neck cancers. Patients are eligible if they are undergoing or scheduled to undergo radiotherapy or chemoradiotherapy in one of the following settings: definitive (primary treatment), adjuvant (post-surgical), or palliative (symptom relief or disease control). The study aims to evaluate treatment effectiveness and monitor side effects across a diverse patient cohort.
Sampling Method: Non-Probability Sample
Enrollment: 915 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Cancer Recurrence | From enrollment to 36 months post-treatment
  The main focus is the probability of recurrence of head and neck cancer after the completion of radiotherapy. This will be assessed at various intervals, specifically at 3, 6, 12, 24, and 36 months post-treatment, using imaging techniques such as PET-CT, MRI, and CT, along with clinical evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Massaccesi, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT06806683/Prot_000.pdf